CLINICAL TRIAL: NCT05284903
Title: Hearing Aid Performance Study for Different Spatial Configurations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: SRF-386
Record Dates: First submitted 2022-03-10; First posted 2022-03-17 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Listening Effort; Noise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Phonak device with activated feature (Other): The clinical investigation is designed to evaluate clinical performances in terms of speech intelligibility and listening effort. The expected benefit is based on clinical relevant differences. This clinical investigation is divided in three parts including Beamformer benefit, Speech Enhancer benefit and Hearing aid benefit (this part will be performed aided).
  Interventions: Other: Beamformer Benefit: Speech intelligibility and Listening effort; Other: Speech Enhancer benefit: Speech intelligibility, Listening effort and Subjective Speech intelligibility; Other: Hearing aid benefit: Speech intelligibility in noise (unaided vs aided condition); Other: Hearing aid benefit: Speech intelligibility in noise (aided condition)
- Comparator: Phonak device with deactivated feature (Other): The comparative testings should be used as reference. The measures will be performed by the same participant group and the same three parts will be evaluated including Beamformer (BF) benefit, Speech Enhancer benefit and Hearing aid benefit. The reference will be performed without these features or with different settings of these features. In case of the Hearing aid benefit, the reference is an unaided fitting.
  Interventions: Other: Beamformer Benefit: Speech intelligibility and Listening effort; Other: Speech Enhancer benefit: Speech intelligibility, Listening effort and Subjective Speech intelligibility; Other: Hearing aid benefit: Speech intelligibility in noise (unaided vs aided condition); Other: Hearing aid benefit: Speech intelligibility in noise (aided condition)

INTERVENTIONS:
Other: Beamformer Benefit: Speech intelligibility and Listening effort — Confirm the improvement in terms of speech intelligibility (measured by OLSA, Oldenburg Sentence Test) and the reduction in terms of listening effort (measured by ACALES) of the I-BF (investigational Beamformer) compared to the R-BF (reference Beamformer), when speech is not coming from the front.
Other: Speech Enhancer benefit: Speech intelligibility, Listening effort and Subjective Speech intelligibility — Confirm the improvement in terms of speech intelligibility (measured by Oldenburg Sentence test) and the reduction in terms of listening effort (measured by ACALES) when the Speech Enhancer is on (SE ON) compared to Speech Enhancer is off (SE OFF) for distant speech or speech from adjacent room.
  Confirm the improvement in terms of subjective level to follow a conversation in quiet when SE ON compared to SE OFF for distant speech or speech from adjacent room. Measured by a subjective assessment.
Other: Hearing aid benefit: Speech intelligibility in noise (unaided vs aided condition) — Confirm the improvement in terms of speech intelligibility (measured by OLSA) in noise with the investigational device (aided condition) compared to the unaided condition.
Other: Hearing aid benefit: Speech intelligibility in noise (aided condition) — Confirm the improvement in terms of speech intelligibility (measured by OLSA) with the Reference binaural beamformer compared to the fixed directional.

SUMMARY:
This clinical investigation will extend the evaluation of perception of speech in different listening environments with hearing aids available on the market (from Phonak). The clinical investigation is divided in three parts addressing different challenges met by hearing aid users.

DETAILED DESCRIPTION:
Hearing aids are designed to amplify and transmit sound to compensate for impaired hearing. The main objective of this medical device is to improve the perception of speech, which can be defined among many attributes by intelligibility or listening effort. Evaluating the performance of the hearing aid or different features reasonably assumes that the talker location should be in front and close of the hearing aid user. However, listening situations in daily life might show much more variability regarding the spatial configuration of the talker, listener and noise sources.

This investigation is designed to extend the evaluation of hearing aid features to different spatial configuration and also to evaluate the benefit of the investigational device. The investigational device is European conformity (CE) marked and will be used within its defined use and on the intended population. The investigation is divided into three independent parts:

* Beamformer (BF) benefit: the first part of the study will evaluate the effect of a wider beamformer on intelligibility and listening effort for a speech-in-noise condition when the talker is not in front of the listener in comparison to a narrower beamformer,
* Speech Enhancer benefit: the second part of the study will evaluate the effect of the Speech Enhancer algorithm on distant speech in quiet and when speech in quiet is coming from an adjacent room with different measures such as listening effort, objective and subjective speech intelligibility,
* Hearing aid benefit: the third part of the study will evaluate the benefit provided by amplification with a speech-in-noise test where the talker is in front and close to the hearing aid user

ELIGIBILITY:
Inclusion Criteria:

* Experienced (minimum use duration 6 months)
* Adult (minimum age: 18 years) hearing aid users,
* Written and spoken German,
* Ability to understand instruction,
* Ability to describe listening experiences,
* Ability to attend to the appointments,
* Healthy outer ear,
* Hearing loss within the fitting ranges of the investigational product,
* Informed consent as documented by signature.

Exclusion Criteria:

* Clinical contraindications deformity of the ear (closed ear canal or absence of pinna),
* Known hypersensitivity or allergy,
* Not willing to wear the hearing aid,
* Fluctuating hearing that could influence the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Speech reception threshold (SRT) for Beamformer Benefit (Oldenburg Sentence Test) | At the test and retest appointment, maximum duration of the test/retest is 120 minutes
  The measure of the speech reception threshold (SRT) is a procedure to evaluate the speech intelligibility in different listening conditions. The SRT in noise is defined as the signal-to-noise ratio (SNR) needed to understand 50% of the presented sentences. The SNR is adapted based on the intelligibility score of the previous sentence. The SRT will be measured with the Oldenburg Sentence Test (OLSA), which is a standard speech intelligibility test in German. The OLSA test uses nonsense sentences with equivalent difficulty.

SECONDARY OUTCOMES:
Listening Effort for Beamformer Benefit (ACALES) | At the test and retest appointment, maximum duration of the test/retest is 120 minutes
  The ACALES will be used to determine listening effort in different situations. Speech stimuli (OLSA sentences) are either presented at different levels in a background noise with fixed level or at different distances from the listener in a quiet environment. This creates different SNRs (speech levels at the position of the listener). The listening effort is subjectively rated on a predefined 13-point categorical scale with varying difficulties (SNRs or talker distance), 1= "no effort", 7 = "moderate effort" to 13 = "extreme effort". ACALES adaptively chooses the SNRs or talker distances for each presentation on the basis of previous ratings.
Listening effort for SE benefit (ACALES) | At the test appointment, maximum duration of the test is 120 minutes
  The ACALES will be used to determine listening effort in different situations. The ACALES will be repeated for 3 distances and 2 conditions (SE Off vs On). The outcome is a rating on a 13 points scale, as the difficulty is fixed by the distance now.
Speech Intelligibility for SE benefit (Oldenburg Sentence Test) | At the test and retest appointment, maximum duration of the test/retest is 120 minutes
  The measure of the speech perception in % is an alternative procedure to evaluate the speech intelligibility in different listening conditions. The Speech perception is defined as % correct words out of a sentence list of 20 sentences. Initially an individual presentation level is measured using adaptive procedure to determine the level necessary to understand 50% of all presented words. Afterwards the correct word score can be obtained using this individual presentation level (reduced by 1 dB) by calculating the ratio of correct words by the number of total words.
Subjective Perception, Subjective Assessment for SE benefit (Questionnaire) | At the test and retest appointment, maximum duration of the test/retest is 120 minutes
  A subjective assessment will be used to determine the subjective perception. For this purpose, a novel is either read by the tester aloud (with soft voice) or presented by a loudspeaker in a reverberant room in three different distances (2m, 4m, 8m) and in an adjacent room with door left ajar.
  The subject rates his/her perception of the presented real and recorded speech using a questionnaire on the dimensions "loudness, listening effort and speech intelligibility". The subjects will rate the perception on the same scale (1- 100%) for both tested conditions (SE Off and SE On) with pencils with different colors to get either absolute and relative ratings.
Speech reception threshold (SRT) for Hearing Aid Benefit (Oldenburg Sentence Test) | At the test appointment, maximum duration of the test is 120 minutes
  The measure of the speech reception threshold (SRT) is a procedure to evaluate the speech intelligibility in different listening conditions. The SRT will be measured with the Oldenburg Sentence Test (OLSA), which is a standard speech intelligibility test in German. SRTs are measured in 3 conditions: unaided, aided with fixed directional and aided with stereo zoom.

CONTACTS AND LOCATIONS:
Locations (1):
- Hörzentrum Oldenburg gGmbH, Oldenburg, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: New implementation of directional beamforming configurations shows improved speech understanding and reduced listening effort — https://www.phonak.com/content/dam/phonak/en/evidence-library/field-studies/PH_FieldStudyNews_LumityDirectionalBeamforming_210x297_EN_028-2475-02_V1-00.pdf

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT05284903/Prot_SAP_000.pdf